CLINICAL TRIAL: NCT05352516
Title: A Randomized, Double-Blind, International Multicentre, Parallel-Controlled Phase III Clinical Study to Evaluate Recombinant Anti-RANKL Human Monoclonal Antibody Injection (HLX14) Versus Denosumab Injection (Prolia®) in Postmenopausal Women With Osteoporosis at High Risk of Fracture
Brief Title: A Study to Evaluate the Efficacy and Safety of HLX14 vs. Denosumab Prolia® in Postmenopausal Women With Osteoporosis at High Risk of Fracture
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX14-002-PMOP301
Record Dates: First submitted 2022-04-23; First posted 2022-04-28 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-07

CONDITIONS: Postmenopausal
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Intervention Model Description: Parallel-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Biological: HLX14
- Control group (Active Comparator)
  Interventions: Biological: Prolia®

INTERVENTIONS:
Biological: HLX14 — Subjects will receive a total of 3 doses of subcutaneous injection of HLX14 (once every 6 months (Q6M)).
  Treatment period 1: D1-D364, subjects will receive subcutaneous injection of HLX14 60mg on D1 and D183.
  Treatment period 2: D365-D546, on D365, subjects will be continue with a third dose of HLX14.
  Arms: Treatment group
Biological: Prolia® — Subjects will receive a total of 3 doses of subcutaneous injection of HLX14 or Prolia® (once every 6 months (Q6M)).
  Treatment period 1: D1-D364, subjects will receive subcutaneous injection of Prolia® 60mg on D1 and D183.
  Treatment period 2: D365-D546, on D365, subjects in the Prolia® arm will be re-randomized 1:1 to either continue with a third dose of Prolia® or transition to HLX14 and receive a single dose of HLX14.
  Arms: Control group

SUMMARY:
This is a randomized, double-blind, international multicentre, parallel-controlled phase III clinical study.

The study plans to enroll 478 postmenopausal women with osteoporosis at high risk of fracture, whom will be randomized at 1:1 to either the experiment group (HLX14) or the control group (Prolia®) based on stratification factors (BMI (< 25, 25-30, > 30) and geographic region (Asian or non-Asian)).

The study includes screening period (28 days), treatment period (total 546 days, contain treatment period 1: D1-D364, treatment period 2: D365-D546), and an end-of-study visit (D547).

DETAILED DESCRIPTION:
* Screening period: From Day -28 to -1, all female with postmenopausal osteoporosis subjects at high risk of fracture sign the informed consent form (ICF) and undergo relevant tests. Those who meet the inclusion criteria and do not meet the exclusion criteria will be randomly assigned into either experiment group (HLX14) or control group (Prolia®) at 1:1 and then enter the treatment period. Vitamin D and calcium supplementation is allowed during the screening period.
* Treatment period: Subjects will receive a total of 3 doses of subcutaneous injection of HLX14 or Prolia® (once every 6 months (Q6M)).

Treatment period 1: D1-D364, subjects will receive subcutaneous injection of HLX14 or Prolia® 60mg on D1 and D183.

Treatment period 2: D365-D546, on D365, subjects in the Prolia® arm will be re-randomized 1:1 to either continue with a third dose of Prolia® or transition to HLX14 and receive a single dose of HLX14. Subjects in the HLX14 arm will be continue with a third dose of HLX14.

* During the treatment period, subjects should taking at least 1000 mg of calcium daily and at least 400 IU of vitamin D daily until the end of study. (Dose will be adjusted by the investigator based on serum calcium)
* End-of-study visit: The end-of-study visit will be conducted on D547 of the study or premature withdrawal. Only serious adverse events related to the investigational product will be recorded thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory postmenopausal women with osteoporosis aged 60-90 years (both inclusive);
2. Postmenopausal, defined as > 2 years of menopause, i.e., > 2 years of spontaneous amenorrhea or > 2 years after bilateral oophorectomy;
3. Bone mineral density (BMD) T-score between -2.5 and -4.0 at the lumbar spine or total hip, i.e., -4.0 < T-score ≤ -2.5, as assessed by the central imaging vendor at the time of screening, based on dual-energy x-ray absorptiometry (DXA) scans;
4. At least 2 vertebrae in the L1-L4 region of lumbar spine and at least one hip are evaluable by DXA, assessed by the central imaging

Exclusion criteria:

1. Diseases that may affect bone metabolism;
2. Thyroid disorders;
3. With serious primary diseases in the cardiovascular, cerebrovascular, or hematopoietic system;
4. Subjects with rheumatoid arthritis or ankylosing spondylitis;
5. Malabsorption syndrome or various gastrointestinal disorders associated with malabsorption;
6. Severe renal impairment due to renal disease with a glomerular filtration rate < 30 mL/min;
7. Hepatic diseases;
8. With serious primary diseases in the cardiovascular, cerebrovascular, or hematopoietic system judged by investigator;
9. Positive for human immunodeficiency virus (HIV) antibody;
10. Vitamin D deficiency;
11. Abnormal serum calcium;
12. Oral and dental diseases;
13. Active or uncontrolled infection requiring systemic therapy within 2 weeks prior to first dose;
14. Type 1 diabetic patients, or type 2 diabetic patients who have poor blood glucose control or are treated with insulin, glucagon-like peptide-1 (GLP-1), thiazolidinediones, SGLT2 inhibitors, etc;
15. Participating in clinical trials of other medical devices or drugs or reaching less than 30 days or 5 half-lives after the last visit in the clinical trials of other medical devices or drugs (non-bone metabolism related drugs) (whichever is longer, calculated from the date of ICF signing). Bone metabolism related drugs should comply with the corresponding prohibition time limit, and anti-osteoporosis drugs should be excluded. Those who have failed in the screening period of other clinical trials but have not yet been treated with drugs/clinical devices can be included in this study;
16. Having received Denosumab and its biosimilars, or Romosozumab and its biosimilars, cathepsin K inhibitor therapy prior to randomization;
17. Having received the following osteoporosis treatments, or medications that affect bone metabolism or any herbal medications:

1) Use of bisphosphonates(oral or intravenous) ,fluoride and strontium prior to randomization.

2) Use of parathyroid hormone (PTH) or PTH analogues, such as teriparatide, within 12 months prior to randomization.

3) Use of systemic hormone replacement therapy (HRT), selective estrogen receptor modulators, tibolone, anabolic hormones, testosterone, androgens, gonadotropin releasing hormone agonists, adrenocorticotropic hormone, within 12 months prior to randomization.

4) Use of calcitonin, calcitriol, alfacalcidol and vitamin D analogues within 12 months prior to randomization: 5) Use of any of the following within 3 months prior to randomization: heparin, warfarin, anticonvulsants (except benzodiazepines), systemic use of ketoconazole, cinacalcet, aluminum, lithium, protease inhibitors, methotrexate, and oral or parenteral glucocorticoids (≥ 5 mg/day prednisone daily or equivalent for > 10 days).

6) Use of any herbal medications within 2 weeks (If the herbal medications contain the above components that affect bone metabolism, should follow the corresponding elution period of bone metabolism components);

18. Subjects with a history or presence of hip fracture or .prevalent vertebral (any severe or more than 2 moderate prevalent vertebral fractures);

19. Subjects in active healing fracture in the opinion of the investigator;

20. Subjects at very high risk of fracture who must be treated immediately with an active drug in the opinion of the investigator;

21. Known allergic to the drugs listed in the study protocol, including a history of allergy to denosumab, any recombinant protein drugs, or any ingredients used in HLX14 or Prolia®;

22. With a history and presence of smoking, except for the following suituation:

1. non-smokers (A history of never smoking > 5 cigarettes/day and not smoking at all for at least the last 2 years prior to screening process)
2. light smokers (with smoking habit <5 cigarettes/day, smoking period <10 years. Light smokers should have not smoked more than 1 cigarette in the week before starting the medical screening process)

23. With a history of drug or alcohol abuse, and with evidence of alcohol or drug abuse within 12 months;

24. Various physical or psychiatric disorders or laboratory abnormalities which, in the opinion of the investigator, will prevent the subject from completing the study or interfere with the interpretation of study results. Or the subjects presenting other factors not suitable for participation in the opinion of the investigator.

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint | 52 Weeks
  Percent change from baseline in BMD at the lumbar spine to Week 52 (D365) (assessed by the central imaging).
  Note: The percent change in BMD is calculated as: (Test value - Baseline value) / (Baseline Value) × 100%
Primary pharmacodynamic endpoint | 26 Weeks
  Area under the effect-time curve for percent change from baseline of serum type I collagen C-telopeptide (s-CTX) from 0 to Week 26 (D183) (AUEC0-26W)

SECONDARY OUTCOMES:
Secondary efficacy endpoint | 78 Weeks
  1. Percent change from baseline in BMD at the lumbar spine to Week 26 (D183), Week 52 (D365),Week78 (D547) (assessed by investigator).
  2. Fracture rate from baseline to Week 52 (D365), Week 78 (D547).
  3. Percent change in BMD at lumbar spine from baseline to Week 26 (D183), Week 78 (D547) (assessed by the central imaging).
  4. Percent change in BMD at total hip from baseline to Week 26 (D183), Week 52 (D365) and Week 78 (D547) (assessed by the central imaging and investigator).
  5. Percent change in BMD at the femoral neck from baseline to Week 26 (D183), Week 52 (D365) and Week 78 (D547) (assessed by the central imaging and investigator).
  Note: Fracture rate=(number of patients with new fractures/total number of patients)*100% The percent change in BMD is calculated as (test value - baseline value) ÷ (baseline value) × 100%
Secondary pharmacodynamic endpoint | 78 Weeks
  1. Relative percent change in serum type I collagen C-telopeptide (s-CTX) from baseline to D15, D29, D57, D92, D106, D134, D162, D183 (within 7 days prior to the second dose), D274, D365 (within 7 days prior to the third dose), and D547 (at the end-of-study visit).
  2. Relative percent changes in serum procollagen type I N propeptide (s-P1NP) from baseline to D15, D29, D57, D92, D106, D134, D162, D183 (within 7 days prior to the second dose), D274, D365 (within 7 days prior to the third dose) and D547 (at the end-of-study visit).
  The relative percent change is calculated as: (Test value at timepoints evaluated - Baseline value) / (Baseline value) × 100%

CONTACTS AND LOCATIONS:
Locations (38):
- China (38):
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Inner Mongolia Baogang hospital, Baotou, Inner Mongolia
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Ruian People's Hospital, Rui'an, Jiangxi
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Beijing BOAI Hospital, Beijing
  - Beijing Hospital, Beijing
  - Beijing Jishuitan Hospital, Beijing
  - BeiJing PINGGU Hospital, Beijing
  - The Third Xiangya Hospital of Central South University, Changsha
  - Changzhou NO.2 People's Hospital, Changzhou
  - West China Hospital of Sichuan University, Chengdu
  - Chongqing University three Gorges Hospital, Chongqing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Department of Geriatrics, Guangzhou First People's Hospital, Guangzhou
  - Guangzhou First People's Hospital, Guangzhou
  - The First Affiliated Hospital of USTC Anhui Provincial Hospital, Hefei
  - Qilu Hospital of Shandong University, Jinan
  - Shandong Provincial Hospital, Jinan
  - Affiliated Hospital of Jining Medical University, Jining
  - The Third People's Hospital of Yunnan Province, Kunming
  - Henan Luoyang Orthopedic Hospital, Luoyang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Jiangxi Provincial People's Hospital, Nanchang
  - Nanchang Hongdu Hospital of traditional Chinese Medicine, Nanchang
  - Nanchang Third Hospital, Nanchang
  - Pingxiang Peoples's Hospital, Pingxiang
  - Suining Central Hospital, Suining
  - First Hospital of Shanxi Medical University, Taiyuan
  - Second hospital of Shanxi Medical University, Taiyuan
  - Tianjin First Central Hospital, Tianjin
  - Weifang People's Hospital, Weifang
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of science and technology, Wuhan
  - Honghui Hospital,Xi'an Jiaotong University, Xi'an

IPD SHARING:
Plan to Share IPD: No